CLINICAL TRIAL: NCT03530059
Title: Feasibility at Home of a Rehabilitation Program Before Thoracic Surgery, for Pulmonary Parenchyma Exeresis
Brief Title: Fast-Track Rehabilitation
Acronym: FTR
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.300; 2017-A02697-46 (Other: ID RCB)
Record Dates: First submitted 2018-02-15; First posted 2018-05-21 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Respiratory Disease; Thoracic Surgery; Lung Cancer
Keywords: Home-based training program
MeSH Terms: conditions — Respiration Disorders; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Home-based rehabilitation — Observational study

SUMMARY:
This study is a prospective observational study which aim to evaluate the feasibility of a total and systematic home respiratory rehabilitation training program in patients who will undergo thoracic surgery, and otherwise tend to define failure reasons.

DETAILED DESCRIPTION:
The aim of this clinical trial is to identify the determining factors which impact a preoperative home respiratory rehabilitation training program success. This success is determined by complete achievement of the program (100%) by the patient.

This rehabilitation program is composed by 4 items:

* Adapted physical activity : 3 averaging cyclo ergometer or physical activity seances per week (25%)
* Physiotherapy sessions : 8 seances with a physical therapist (25%)
* Smokers : Set up of a program to help give up smoking if active smoker (25%)
* Dietetics : If unintentionally weight loss (>5% total weight in 1 month or >10% in 6 months) or BMI<21 , nutritional assessment is conducted and dietetic program is initiated(25%)

Secondary objectives are :

* Assessment of postoperative event onset (30 days) (atelectasis, fibro-aspiration, time spent in resuscitation unit, intubation, revision surgery).
* Link assessment of 100% program success and at least one complication onset.
* Cost assessment of preoperative rehabilitation program
* Evaluation of mean hospitalisation duration post surgery (30 days)
* Average cost assessment of hospitalisation stay per patient.

This study will include 50 patients over 18 years old, addressed to the home heath care provider AGIR à Dom, for rehabilitation before pulmonary parenchyma exeresis.

Patients must perform at least 2 items of rehabilitation program previously described.

This program is an initiative of a pulmonologist or a thoracic surgeon, who include the patient when the date of surgery is scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need a respiratory rehabilitation before thoracic surgery for lung resection.
* Patients addressed to the home heath care provider "AGIR à Dom",
* Patients must perform at least 2 items of rehabilitation program (Adapted physical activity, Diet, Physiologist, Smoking)

Exclusion Criteria:

* Patients who participate to another interventional research that may impact this study.
* Patients unable to get involved to the training program, depending to the investigator's appreciation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * All patients over 18 years old referred by a pulmonologist or a thoracic surgeon for a thoracic surgery of pulmonary lobe or lung removal.
  * Be able physically and be enthousiastic to engage a home-training respiratory program.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-07-21 (Actual)

PRIMARY OUTCOMES:
Completion (yes/no) of the home-training program based on 4 items: tobacco, dietary, physical activity and physiotherapy before thoracic surgery | from date of inclusion until the end of hospitalisation for thoracic surgery, assessed up to 6 months
  Completion (yes/no) of the home-training program based on 4 items: tobacco, dietary, physical activity and physiotherapy before thoracic surgery :
  * Tobacco: measure of tobacco consumption (self-report)
  * Dietary: body mass
  * Physical activity: number of physical activity sessions
  * Physiotherapy: number of physical therapy sessions

SECONDARY OUTCOMES:
Post operative event number | 30 days
  Post operative event number
Rehabilitation program costs | from date of inclusion until the beginning of hospitalisation for thoracic surgery, assessed up to 6 months
  Rehabilitation program costs before surgery for the 4 program rehabilitation items
Hospitalisation duration | from the beginning until the end of hospitalisation for thoracic surgery, assessed up to 3 months
  Hospitalisation duration in days per unit
Total hospitalisation cost | from the beginning until the end of hospitalisation for thoracic surgery, assessed up to 3 months
  Total hospitalisation cost per patient = sum for all unit

CONTACTS AND LOCATIONS:
Overall Officials: François ARBIB, MD-PhD, Principal Investigator — CHUGA
Locations (5):
- France (5):
  - Centre Medivallee, Saint-Ismier, ZI La Batie 35 Allée Du Champrond
  - Maison Medicale Des Cedres, Échirolles
  - GROUPE HOSPITALIER MUTUALISTE INSTITUT de CANCEROLOGIE DANIEL HOLLARD, Grenoble
  - Chu Grenoble Alpes, Grenoble
  - Cabinet de Chirurgie Cardio Vasculaire, Saint-Martin-d'Hères

REFERENCES:
- [Derived] Catho H, Guigard S, Toffart AC, Frey G, Chollier T, Brichon PY, Roux JF, Sakhri L, Bertrand D, Aguirre C, Gorain S, Wuyam B, Arbib F, Borel JC. What are the barriers to the completion of a home-based rehabilitation programme for patients awaiting surgery for lung cancer: a prospective observational study. BMJ Open. 2021 Feb 10;11(2):e041907. doi: 10.1136/bmjopen-2020-041907. PMID 33568371